CLINICAL TRIAL: NCT04295226
Title: Structured Post-stroke Follow-up at Skåne University Hospital in Malmö, Sweden - a Feasibility and Validation Study (SUESIM)
Brief Title: Structured Post-stroke Follow-up in Malmö, Sweden (SUESIM)
Acronym: SUESIM
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Collaborators: The Kamprad Family Foundation for Entrepreneurship, Research & Charity (Other); Clinical Studies Sweden - Forum South (Unknown); Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/1028
Record Dates: First submitted 2019-04-28; First posted 2020-03-04 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Stroke
Keywords: follow-up; post stroke checklist; complications
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants in Structured post-stroke follow-up in Malmö: Consecutive patients with acute ischemic stroke or intracerebral hemorrhage, treated in-hospital at Skåne University Hospital in Malmö and discharged straight to own home.
  The intervention consists of a structured follow-up visit, managed by a stroke nurse, 3 months after stroke followed by a multidisciplinary team rounds resulting in an individual treatment plan for stroke-related health problems, and a final follow-up at 12 months
  Interventions: Other: Structured follow-up after stroke.

INTERVENTIONS:
Other: Structured follow-up after stroke. — Stroke-nurse managed follow-up 3 and 12 months after stroke and multidisciplinary rounds resulting in individual treatment plans for stroke-related health problems.

SUMMARY:
Background Stroke-related medical complications and health problems are common among stroke survivors. Post-stroke Checklist (PSC), developed by an international expert group, and can be used as a clinical tool to identify common and treatable stroke-related health problems. PSC has not been systematically tested in Sweden.

Aims To test the feasibility of a structured and multimodal follow-up model for stroke systematically, to test the validity of the PSC as a screening tool for stroke-related health problems and to study the prevalence of, and changes over time, of stroke-related health problems Study population We plan to include 200 consecutive patients with acute stroke, treated in-hospital at Skåne University Hospital in Malmö and discharged straight to own home.

Procedure The intervention consists of a structured follow-up visit, managed by a stroke nurse, 3 months after stroke followed by a multidisciplinary team rounds resulting in an individual treatment plan for stroke-related health problems, and a final follow-up at 12 months.

Feasibility will be evaluated, as well as burden of stroke-related health problems and interventions prompted by the visits.

Researchers responsible for the study:

Teresa Ullberg, MD, Ph (Postdoctoral researcher) and Hélène Pessah-Rasmussen, MD, PhD, associate professor (PI).

DETAILED DESCRIPTION:
Background Approximately 600 patients with acute stroke are treated in-hospital at Skåne University Hospital in Malmö. Of those, approximately 450 patients can be discharged straight to their own home after hospital stay. Currently, there is no structured follow-up routine for patients with stroke discharged from Skåne University Hospital in Malmö, and Primary care health providers are managing most follow-ups for stroke depending on individual patient needs. Previous research has shown that one in four patients with stroke are not followed up within three months after hospital discharge in Skåne.

Stroke-related medical complications are common both in the acute phase after stroke and in the longer term. Acute medical complications comprise infections, falls and fractures, confusion, deep venous thrombosis and pulmonary embolism, and also epileptic seizures. The risk of medical complications increases with co-morbidity, but can also be a consequence of the stroke itself. Beyond the acute phase, other stroke-related health problems occur in the majority of patients. They comprise fatigue, impaired cognition, low mood, incontinence, sexual impairment, post-stroke pain, spasticity, relational problems, isolation, inadequate secondary preventive treatment and impaired mobility and daily activities. Previous studies have shown that these problems are common and can persist for years post-stroke. Knowledge of how to best organize and manage stroke and stroke-related health problems in the long-term is sparse, even though there are guidelines on some general principles for secondary prevention and rehabilitation.

Post-stroke Checklist (PSC) was developed by an international stroke expert group. It is a simple checklist collecting eleven common stroke-related health problems, and can be used as a clinical tool to identify common and treatable complications to stroke. The feasibility of the 11-items PSC as a screening tool for stroke-related health problems has been tested systematically and it has been considered implementable. Modified versions of PSC are being implemented in different countries.

PSC can be used both by nurses, physicians and other health professions. The National Guidelines for Stroke Care in Sweden from 2018 recommend the use of PSC for stroke follow-up. PSCs use has not been systematically tested in Sweden though and PSC is not yet routinely used. A modified 14-item PSC is recommended by Region Skåne (the county council of Southern Sweden).

Aims The aims of this study are to test the feasibility of a structured and multimodal follow-up model for stroke systematically, as well as to test the validity of the PSC as a screening tool for stroke-related health problems. The study aims further at studying the prevalence, and changes over time, of stroke-related health problems as well as survival, functional outcome following stroke, and patient satisfaction.

Working plan Study design The study design is longitudinal and explorative. This is a feasibility and validation study where the intervention consists of a structured follow-up visit, a multidisciplinary team rounds resulting in an individual treatment plan for stroke-related health problems, and a final follow-up at 12 months. Individual items in PSC will be validated towards routinely used validated tools. The prevalence, and changes over time, of stroke-related health problems will be investigated, as well as survival, functional outcome following stroke, and patient satisfaction. The study takes place in the clinical setting at the stroke unit, using clinical stroke team professional to mimic the normal clinical situation.

Study population We plan to include 200 consecutive patients with acute ischemic stroke or intracerebral hemorrhage, treated in-hospital at Skåne University Hospital in Malmö and discharged straight to own home. The estimated inclusion rate is 3- 5 patients per week, and the estimated time for including 200 patients is one year. Two hundred patients represent 40% of the total population of the 500 patients who can be discharged straight to own home, and are expected to be representable of the population with respect to age, sex, vascular risk and stroke severity. The generalizability of the population will be assessed through comparison to the Swedish Stroke Register.

Procedure for inclusion Eligible patients are identified daily in the stroke ward and included by written informed consent.

Follow-up procedure The three-months visit is managed by a stroke nurse and include the semi-structured PSC interview, additional validated diagnostic tools, secondary prevention status, comorbidity, and functional outcome.

The three-months visit is followed by a multidisciplinary team rounds with stroke physician, stroke nurse, occupational therapist and if needed physiotherapist, speech therapist, dietician, psychologist and/or social worker. The rounds result in an individual treatment recommendation plan that is sent to the family doctor and other relevant instances. The amount and type of referrals and other interventions warranted by the results of the follow-up visits and rounds are recorded.

The 12-months visit is managed by a stroke nurse and include a new semi-structured PSC interview, secondary prevention status, comorbidity, and a met needs assessment. The 12-month visit is followed by a multidisciplinary team rounds leading to referrals and other interventions are if warranted.

Use of other register data Patient baseline characteristics and three- and 12-month data on living conditions and functional level will be obtained from the Swedish Stroke Register (Riksstroke). Mortality at 12 and 18 months will be obtained by linkage to the Swedish Causes of Death register.

Data management, statistical analyses and ethical considerations The database will be built and managed in close cooperation with Clinical Studies Sweden, Forum South. Analyses will be performed on de-identified data after the dataset has been closed.

All statistical analyses will be performed in SPSS. Data will be presented using descriptive statistics and graphs, as well as linear models. Power calculations are not relevant for this study type.

The local Ethics approval committee has approved of the project (Dnr 2017/1028)

ELIGIBILITY:
Inclusion Criteria:

* Acute stroke (ICD-10: ischemic stroke I.63 and intracerebral hemorrhage I.61)
* Discharge to own home

Exclusion Criteria:

* Co-morbidity such as dialysis, active cancer, severe heart failure or severe psychiatric illness or dementia
* Patients with stroke, but who receive in-hospital treatment for another competing diagnosis
* Already included with previous stroke
* Does not want to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with acute stroke, without dementia or other serious comorbidity, that can be discharged straight home. These patients have mild to moderate stroke and can be expected to be able to visit an out-patient clinic for follow-up and to benefit from a structured follow-up visit.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Number of stroke-related health problems | 1 year
  14-item Post-stroke Checklist, PSC, captures 14 stroke-related health problems. Scale ranges from 0-14 problems. We aim to analyse burden of problems as well as individual items.
Number of interventions | 1 year
  Number of new interventions for stroke-related health problems identified with PSC. No scale used, we calculate the number of interventions done.

SECONDARY OUTCOMES:
Time to perform and record the semi-structured Post-Stroke Checklist (PSC) interview (minutes). | 1 year
  Feasibility of the post-stroke checklist-based follow-up. No scale used, only time in minutes.
Ability to complete all Post-Stroke Checklist (PSC) items (yes/no) | 1 year
  Feasibility of the post-stroke checklist-based follow-up. No scale used. Dichotomous variable (yes/no)
Patient satisfaction assessment | 1 year
  Questionnaire on met needs and satisfaction with follow-up. Five dichotomous questions on met needs and satisfaction with follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Skåne university hospital, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ullberg T, Zia E, Petersson J, Norrving B. Doctor's follow-up after stroke in the south of Sweden: An observational study from the Swedish stroke register (Riksstroke). Eur Stroke J. 2016 Jun;1(2):114-121. doi: 10.1177/2396987316650597. Epub 2016 May 19. PMID 31008273
- [Background] Kumar S, Selim MH, Caplan LR. Medical complications after stroke. Lancet Neurol. 2010 Jan;9(1):105-18. doi: 10.1016/S1474-4422(09)70266-2. PMID 20083041
- [Background] Langhorne P, Stott DJ, Robertson L, MacDonald J, Jones L, McAlpine C, Dick F, Taylor GS, Murray G. Medical complications after stroke: a multicenter study. Stroke. 2000 Jun;31(6):1223-9. doi: 10.1161/01.str.31.6.1223. PMID 10835436
- [Background] Ullberg T, Zia E, Petersson J, Norrving B. Perceived Unmet Rehabilitation Needs 1 Year After Stroke: An Observational Study From the Swedish Stroke Register. Stroke. 2016 Feb;47(2):539-41. doi: 10.1161/STROKEAHA.115.011670. Epub 2016 Jan 5. PMID 26732564
- [Background] McKevitt C, Fudge N, Redfern J, Sheldenkar A, Crichton S, Rudd AR, Forster A, Young J, Nazareth I, Silver LE, Rothwell PM, Wolfe CD. Self-reported long-term needs after stroke. Stroke. 2011 May;42(5):1398-403. doi: 10.1161/STROKEAHA.110.598839. Epub 2011 Mar 24. PMID 21441153
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Lancet. 2007 Oct 20;370(9596):1453-7. doi: 10.1016/S0140-6736(07)61602-X. PMID 18064739
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] Murray J, Young J, Forster A, Ashworth R. Developing a primary care-based stroke model: the prevalence of longer-term problems experienced by patients and carers. Br J Gen Pract. 2003 Oct;53(495):803-7. PMID 14601359
- [Background] Philp I, Brainin M, Walker MF, Ward AB, Gillard P, Shields AL, Norrving B; Global Stroke Community Advisory Panel. Development of a poststroke checklist to standardize follow-up care for stroke survivors. J Stroke Cerebrovasc Dis. 2013 Oct;22(7):e173-80. doi: 10.1016/j.jstrokecerebrovasdis.2012.10.016. Epub 2012 Dec 21. PMID 23265778
- [Background] Ward AB, Chen C, Norrving B, Gillard P, Walker MF, Blackburn S, Holloway L, Brainin M, Philp I; Global Stroke Community Advisory Panel (GSCAP). Evaluation of the Post Stroke Checklist: a pilot study in the United Kingdom and Singapore. Int J Stroke. 2014 Oct;9 Suppl A100:76-84. doi: 10.1111/ijs.12291. Epub 2014 Aug 4. PMID 25088427
- [Derived] Mansson K, Soderholm M, Berhin I, Pessah-Rasmussen H, Ullberg T. The Post-Stroke Checklist: longitudinal use in routine clinical practice during first year after stroke. BMC Cardiovasc Disord. 2024 Oct 29;24(1):601. doi: 10.1186/s12872-024-04239-6. PMID 39468444
- See also: Quality register — http://www.Riksstroke.Org/eng/